CLINICAL TRIAL: NCT04108273
Title: Brain Plasticity Underlying Acquisition of New Organizational Skills in Children
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: NYU Langone Health (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: s17-00263; R61MH113663 (NIH)
Record Dates: First submitted 2019-09-26; First posted 2019-09-30 (Actual); Results first posted 2024-08-01 (Actual); Last update posted 2024-08-01 (Actual); Status verified 2024-07

CONDITIONS: ADHD; Attention Deficit Hyperactivity Disorder; Neurodevelopmental Disorders
MeSH Terms: conditions — Attention Deficit Disorder with Hyperactivity; Neurodevelopmental Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- No-Wait (Experimental): Participants with organizational skill difficulties to undergo two magnetic resonance imaging (MRI) sessions: one within 2 weeks prior to OST treatment and one within 2 weeks of completion of the OST treatment.
  Interventions: Behavioral: Organizational Skills Training
- Waitlist (Active Comparator): Participants with organizational skill difficulties to undergo two magnetic resonance imaging (MRI) sessions: one 12 weeks prior to OST treatment and one ~12 weeks after their first scan and before proceeding to OST.
  Interventions: Behavioral: Organizational Skills Training

INTERVENTIONS:
Behavioral: Organizational Skills Training — OST targets three core organizational skills domains - Tracking Assignments, Managing Materials and Time Management - in a program consisting of sessions over 12 weeks, each training lasting about 1 hour, and corresponding 30-60 minute weekly review sessions with the parent and the child, 2-3 days following each training session.

SUMMARY:
Organizational, time management and planning (OTMP) skills deficits are impairing features of developmental disorders, such as Attention Deficit Hyperactive Disorder (ADHD), which compromise school performance and family relations. The manualized Organizational Skills Training program (OST) was designed to target children's specific OTMP deficits. However, the brain mechanisms of treatment-induced changes remain unknown. The current study combines a training intervention (OST) with non-invasive MRI imaging in a pre-/post-design in a randomized two-arm (treatment vs. waitlist) trial to address this question.

ELIGIBILITY:
Inclusion Criteria:

* Age at entry: age ≥ 8.0 and ≤ 11.9 years corresponding to grades 3-5
* Written assent by child and consent by parent or legal guardian
* IQ: Estimated full scale IQ ≥ 85 and language comprehension scores ≥ 8
* Organizational skills deficits defined as elevated (≥ 1SD) pre-treatment Children's Organizational Skills Scales (COSS) Parent Total T-score and at least one COSS Parent Interference item rated as either a 3 or 4 (indicating an above-average level of impairment)
* Must provide adequate MRI data at baseline

Exclusion Criteria:

* Enrolled in a self-contained special education classroom or served by a 1:1 paraprofessional in their classroom
* Absence of signed consent by parent or legal guardian
* Children who dissent regardless of parental permission
* Full scale IQ < 85
* Children with a recent (past 6 months) or current history of neuroleptic treatment or current treatment with psychotropic medications other than stimulants
* Per history (and medical records if needed) medical illness requiring chronic current treatment
* History of intrathecal chemotherapy or focal cranial irradiation
* Premature birth (< 32 weeks estimated gestational age or birth weight < 1500g)
* History of leukomalacia or static encephalopathy, intracerebral hemorrhage beyond grade 2, other specific or focal neurological or metabolic disorder including epilepsy (except for resolved febrile seizures)
* History of traumatic brain injury
* Contraindication for MRI scanning (metal implants, pacemakers, metal foreign bodies or pregnancy)

Ages: 8 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 59 (Actual)
Dates: Start 2019-10-01 (Actual); Primary Completion 2023-06-20 (Actual); Study Completion 2023-08-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Francisco Castellanos, MD, Principal Investigator — New York Langone Health
Locations (1):
- NYU Langone Health, New York, New York, United States

IPD SHARING:
Plan to Share IPD: Yes
De-identified individual participant data will be provided to the NIMH Data Archive (NDA) for sharing to investigators
Supporting Information: Study Protocol, SAP

REFERENCES:
- [Derived] Martinez Agulleiro L, Deng B, Gallagher R, Abikoff HB, Yoncheva Y, Robinson L, Conlon G, Haroon M, Yan CG, Di Martino A, Zhao Y, Castellanos FX. Brain plasticity underlying acquisition of new organizational skills in children: A Rashomon analysis. Front Neuroimaging. 2025 Dec 9;4:1671310. doi: 10.3389/fnimg.2025.1671310. eCollection 2025. PMID 41446359

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | No-Wait | Waitlist
Started | 30 | 29
Completed | 29 | 29
Not Completed | 1 | 0
Not completed — COVID Pandemic | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | No-Wait | Waitlist | Total
Number analyzed (Participants) | 29 | 29 | 58
Age, Continuous [Mean (Standard Deviation); unit: years] | 9.5 (0.949) | 9.4 (0.686) | 9.5 (0.821)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 11 | 11 | 22
  Male | 18 | 18 | 36
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 7 | 3 | 10
  Not Hispanic or Latino | 22 | 26 | 48
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 4 | 4
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 1 | 1
  White | 21 | 15 | 36
  More than one race | 5 | 9 | 14
  Unknown or Not Reported | 3 | 0 | 3
Region of Enrollment [Number; unit: participants]
  United States | 29 | 29 | 58

OUTCOME MEASURES:

1. Primary Outcome: Change in the Intrinsic Functional Connectivity (iFC) Between Dorsal Anterior Cingulate Cortex (dACC) and Default Mode Network Subdivision of the Anterior Ventral Striatum (aVS-DMN)
Description: The iFC between the two regions was measured at both baseline and follow-up by calculating the Fisher Z-transformed correlation between the average time-series of all voxels within each region of interest (positive values indicate increased iFC between the two regions, while negative values indicate decreased iFC). Then, to determine the change in iFC due to the intervention/waitlist period, the iFC between both regions at baseline was subtracted from the iFC between both regions at follow-up. Therefore, this provides a measure of the change in iFC due to the intervention or waitlist period, with positive values indicating an increase in iFC and negative values indicating a decrease in iFC due to the intervention/waitlist period.
Time Frame: baseline MRI, second MRI visit (treatment arm ~14 weeks, waitlist arm ~12 weeks)
Measure: Mean (Standard Deviation); unit: Fisher transformed z values
Arm/Group | No-Wait | Waitlist
Number analyzed (Participants) | 25 | 26
Fisher transformed z values | -0.07 (0.214) | 0.01 (0.196)

2. Primary Outcome: Change in Parent Children's Organizational Skills Scales (COSS-P) Total T-scores Following OST Intervention
Description: The Children's Organizational Skills Scale quantifies how children (ages 8-13) organize their time, materials, and actions to accomplish important tasks at home and school. The Parent report consists of 66 questions, each using a 4-point Likert-type scale (where 1=Hardly ever or never and 4=just about all the time). Scores are normalized to a T-distribution, with a population mean of 50; scores of 60 or above are considered evidence of deficient organizational skills.
Time Frame: baseline, second MRI visit (treatment arm ~14 weeks, waitlist arm ~12 weeks)
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | No-Wait | Waitlist
Number analyzed (Participants) | 26 | 26
scores on a scale | -14.8 (7.61) | -3.5 (5.87)

3. Primary Outcome: Change in the Intrinsic Functional Connectivity (iFC) Between Dorsal Anterior Cingulate Cortex (dACC) and Fronto Parietal Network Subdivision of the Anterior Ventral Striatum (aVS-FP)
Description: as for outcome 1
Time Frame: baseline MRI, second MRI visit (treatment arm ~14 weeks, waitlist arm ~12 weeks)
Measure: Mean (Standard Deviation); unit: Fisher transformed z values
Arm/Group | No-Wait | Waitlist
Number analyzed (Participants) | 25 | 26
Fisher transformed z values | -0.13 (0.213) | -0.1 (0.182)

4. Primary Outcome: Change in the Intrinsic Functional Connectivity (iFC) Between Dorsal Anterior Cingulate Cortex (dACC) and Limbic Network Subdivision of the Anterior Ventral Striatum (aVS-LIM)
Description: as for outcome 1
Time Frame: baseline MRI, second MRI visit (treatment arm ~14 weeks, waitlist arm ~12 weeks)
Measure: Mean (Standard Deviation); unit: Fisher transformed z values
Arm/Group | No-Wait | Waitlist
Number analyzed (Participants) | 25 | 26
Fisher transformed z values | 0.003 (0.176) | 0.0003 (0.165)

ADVERSE EVENTS:
Time Frame: Participants in the active arm were assessed during the period they received the intervention (i.e., since baseline until the last visit, up to 14 weeks). Participants in the waitlist arm were not assessed for adverse events.
Arm/Group | No-Wait | Waitlist
All-Cause Mortality (participants affected / at risk) | 0/29 | 0/29
Serious Adverse Events (participants affected / at risk) | 0/29 | 0/29
Other Adverse Events (participants affected / at risk) | 0/29 | 0/29

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2023-05-30): https://cdn.clinicaltrials.gov/large-docs/73/NCT04108273/Prot_SAP_000.pdf